CLINICAL TRIAL: NCT00219765
Title: Phase I/II Trial to Study the Dose, Tolerability and the Effectiveness of Imatinib in Combination With Daunorubicine and Cytarabine for Patients With Chronic Myelogenous Leukemia in Myeloid Acute Phase
Brief Title: Safety and Efficacy of Imatinib in Combination With High Dose Chemotherapy for Acute Phase Chronic Myelogenous Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010495; CSTI571AFR01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; Acute Phase; Imatinib mesylate; Cytarabine; Daunorubicine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Cytarabine; Daunorubicin

INTERVENTIONS:
Drug: Imatinib mesylate 600 mg
Drug: Cytarabine
Drug: Daunorubicine

SUMMARY:
The aim of this phase I/II trial is to determine the dose of daunorubicine to be associated with cytarabine and Imatinib for induction therapy in patients with chronic myelogenous leukemia in myeloid acute phase.

DETAILED DESCRIPTION:
Study design Imatinib: starting at day -3: 600mg/day; continuous administration In combination with cytarabine: continuous iv/24h: 100mg/m² ; 7 days and daunorubicine: 4 levels

level 1: 0

level 2: 15mg/m² ; 3 days

level 3: 30mg/m² ; 3 days

level 4: 45mg/m² ; 3 days

ELIGIBILITY:
Inclusion Criteria:

* CML Ph+ (assessed by cytogenetic or FISH)
* Acute phase with ≥ 20% bone marrow blasts (M0 to M6 , excluding M3)
* Age ≥ 18 year at inclusion
* PS grade 0 to 2 (ECOG)
* Adequate and organ function, defined as the following: total bilirubin <1.5x uln, sgpt <3x uln, creatinine <1.5x uln.
* Informed consent signed up

Exclusion Criteria:

* active malignancy other than CML or non-melanoma cancer of the skin
* current treatment with another investigational agent
* patients with grade 3/4 cardiac disease or any other serious concurrent medical condition.
* patients who are pregnant or nursing. All patients of childbearing potential must practice effective methods of contraception while on study.
* patients with mental illness or other condition precluding their ability to give informed consent or to comply with study requirements patients with performans status 3-4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-05; Study Completion 2006-01

PRIMARY OUTCOMES:
To assess the tolerability and the effectiveness of imatinib in combination with daunorubicine and cytarabine and to determine the recommended dose of daunorubicine to be associated with cytarabine

SECONDARY OUTCOMES:
- To evaluate the survival without progression, the survival without event, the overall survival, the hematologic, cytogenetic and molecular responses at various check points.
- To evaluate duration of responses and failure to respond

CONTACTS AND LOCATIONS:
Overall Officials: François GUILHOT, MD, Study Chair — Department of Oncology hematology and Cell therapy, University Hospital , 86021 Poitiers - FRANCE
Locations (1):
- University Hospital, Poitiers, France

REFERENCES:
- [Derived] Rousselot P, Cony-Makhoul P, Nicolini F, Mahon FX, Berthou C, Rea D, Reiffers J, Bornand A, Saint-Jean O, Guilhot J, Guilhot F; French Intergroup For Chronic Myelogenous Leukemia (Fi-LMC). Long-term safety and efficacy of imatinib mesylate (Gleevec(R)) in elderly patients with chronic phase chronic myelogenous leukemia: results of the AFR04 study. Am J Hematol. 2013 Jan;88(1):1-4. doi: 10.1002/ajh.23330. Epub 2012 Sep 17. PMID 22987312
- [Derived] Deau B, Nicolini FE, Guilhot J, Huguet F, Guerci A, Legros L, Pautas C, Berthou C, Guyotat D, Cony-Makhoul P, Gardembas M, Michallet M, Hayette S, Cayuela JM, Weiss IR, Rea D, Castaigne S, Mahon FX, Guilhot F, Rousselot P. The addition of daunorubicin to imatinib mesylate in combination with cytarabine improves the response rate and the survival of patients with myeloid blast crisis chronic myelogenous leukemia (AFR01 study). Leuk Res. 2011 Jun;35(6):777-82. doi: 10.1016/j.leukres.2010.11.004. Epub 2010 Dec 10. PMID 21145590